CLINICAL TRIAL: NCT05043935
Title: The Effect of Leukocyte and Platelet-rich Fibrin With Antimicrobial Photodynamic Therapy in Treatment of Aggressive Periodontitis Patients: A Randomized Controlled Clinical Trial
Brief Title: The Effect of Leukocyte and Platelet-rich Fibrin With Antimicrobial Photodynamic Therapy in Aggressive Periodontitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Dalia Rasheed Issa, principle investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: waiting
Record Dates: First submitted 2021-08-20; First posted 2021-09-14 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: L-PRF; Photodynamic Therapy; Aggressive Periodontitis
MeSH Terms: conditions — Aggressive Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-PRF with antimicrobial photodynamic therapy (Experimental): Application of L-PRF with antimicrobial photodynamic therapy in the defect
  Interventions: Procedure: L-PRF with antimicrobial photodynamic therapy
- antimicrobial photodynamic therapy (Active Comparator): Application antimicrobial photodynamic therapy in the defect
  Interventions: Procedure: antimicrobial photodynamic therapy without L-PRF

INTERVENTIONS:
Procedure: L-PRF with antimicrobial photodynamic therapy — Application of L-PRF with antimicrobial photodynamic therapy in the defect
  Arms: L-PRF with antimicrobial photodynamic therapy
Procedure: antimicrobial photodynamic therapy without L-PRF — application of antimicrobial photodynamic therapy without L-PRF in the defect
  Arms: antimicrobial photodynamic therapy

SUMMARY:
Antimicrobial photodynamic therapy (aPDT) is associated with photosensitizing agents which promote the generation of free radicals and singlet oxygen, which are cytotoxic to certain bacteria. Leukocyte and platelet-rich fibrin (L-PRF) has been used extensively in the treatment of intrabony defects and achieved excellent results. It acts as an immune regulation node with inflammation control abilities, including a slow continuous release of growth factors which stimulates periodontal regeneration. The aim of this study is to evaluate the adjunctive effects of aPDT with and without L-PRF in aggressive periodontitis patients.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* non- smoker,
* not received any periodontal treatment within the last 6 months,
* no antibiotics, anti- inflammatory drugs or any other medication taken within the last 6 months

Exclusion Criteria:

* any systemic disease that might influence the prognosis of periodontal disease and outcome of the treatment,
* any medical condition that required antibiotic prophylaxis before the treatment,
* smoking,
* pregnancy and lactation,
* ingestion of antibiotics, anti-inflammatory drugs or any other medication during the study period,
* any physical limitations or restrictions that might preclude normal oral hygiene procedures.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation and measurements of the defect in millimeters | 9 months
  Changes in clinical measurements in millimeters after application of antimicrobial photodynamic therapy with and without L-PRF
Radiographic evaluation and measurements of the defect in millimeters | 9 months
  Changes in bone formation in millimeters after application of antimicrobial photodynamic therapy with and without L-PRF

CONTACTS AND LOCATIONS:
Overall Officials: Dalia R Issa, PhD, Principal Investigator — Kafrelsheikh University
Locations (1):
- Faculty of Dentistry, Kafrelsheikh University, Kafr ash Shaykh, Egypt